CLINICAL TRIAL: NCT04418479
Title: Clopidogrel Versus Aspirin Monotherapy After Percutaneous Coronary Intervention and Standard Dual Antiplatelet Therapy in Patients At High Risk for Recurrent Ischemic Events
Brief Title: SMart Angioplasty Research Team: CHoice of Optimal Anti-Thrombotic Strategy in Patients Undergoing Implantation of Coronary Drug-Eluting Stents 3
Acronym: SMART-CHOICE3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joo-Yong Hahn (Other)
Responsible Party: Sponsor-Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOICE-3
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Antiplatelet Therapy; Complex Coronary Lesion; Aspirin; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, two-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin monotherapy arm (Active Comparator): Patients will receive 100 mg of aspirin once daily.
  Interventions: Drug: Aspirin
- Clopidogrel monotherapy arm (Experimental): Patients will receive 75 mg of clopidogrel once daily.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — Randomization will be performed 1:1 between clopidogrel and aspirin monotherapy in patients who completed standard duration of dual antiplatelet therapy (DAPT) and who were at high risk for recurrent ischemic events after percutaneous coronary intervention (PCI) with drug-eluting stent (DES).
  This group will be taken aspirin 100 mg once daily during the study period.
  Other Names: Aspirin monotherapy
  Arms: Aspirin monotherapy arm
Drug: Clopidogrel — Randomization will be performed 1:1 between clopidogrel and aspirin monotherapy in patients who completed standard duration of dual antiplatelet therapy (DAPT) and who were at high risk for recurrent ischemic events after percutaneous coronary intervention (PCI) with drug-eluting stent (DES).
  This group will be taken clopidogrel 75 mg once daily during the study period.
  Other Names: Clopidogrel monotherapy
  Arms: Clopidogrel monotherapy arm

SUMMARY:
This study is a prospective, open-label, two-arm, randomized multicenter trial to compare the efficacy and safety of clopidogrel versus aspirin monotherapy beyond the standard duration of dual antiplatelet therapy (DAPT) (more than 12 months for myocardial infarction [MI] and more than 6 months for non-MI) after percutaneous coronary intervention (PCI) in patients at high risk of recurrent ischemic events.

DETAILED DESCRIPTION:
After the introduction of the second-generation drug-eluting stents (DES), the rates of device-related failure or target lesion failure such as restenosis and stent thrombosis has been markedly decreased, compared with the era of bare-metal stents or first-generation DES. Nevertheless, the risk of ischemic events including very late stent thrombosis after percutaneous coronary intervention (PCI) has still remained even though the use of second-generation DES. In this regard, the ACC (American College of Cardiology)/AHA (American Heart Association) and ESC (European Society of Cardiology) guidelines recommended that dual antiplatelet therapy (DAPT) should be considered for 12 months or longer in patients presented with acute coronary syndrome (ACS) and for 6 months or longer in patients presented with stable ischemic heart disease (SIHD) after PCI with DES. In particular, patients presented with a high risk of ischemic events such as diabetes mellitus, myocardial infarction, or complex coronary lesions were associated with significantly increased future recurrent ischemic events after PCI with DES. In addition, maintenance of DAPT for 12 months or longer has been shown to reduce the recurrence of ischemic events up to 44% in patients treated with PCI for complex coronary artery lesion; therefore the current guideline recommended that prolonged DAPT might be considered when performing complex PCI. However, prolonged DAPT increases bleeding risk and cost. Endoscopic, dental, and surgical procedures are often delayed due to prolonged DAPT, which may affect the patient's quality of life. Therefore, to determine the optimal or minimal necessary duration of DAPT is very important.

The other important issue is that which antiplatelet agent is more appropriate after DAPT. Aspirin monotherapy has been recommended traditionally. However, there is no randomized comparison study between aspirin monotherapy versus clopidogrel monotherapy after DAPT in patients undergoing PCI with DES. Furthermore, clopidogrel is also actively used as a monotherapy after DAPT in real-world practice. In CAPRIE (clopidogrel versus aspirin in patients at risk of ischemic events) trial, clopidogrel showed a superior efficacy in preventing ischemic events compared with aspirin. Moreover, the incidence of gastrointestinal bleeding was significantly lower with clopidogrel than with aspirin. Clopidogrel monotherapy can reduce ischemic events and bleeding risk compared with aspirin monotherapy.

Therefore, the purpose of the SMART-CHOICE 3 (SMart Angioplasty Research Team: CHoice of Optimal Anti-Thrombotic Strategy in Patients Undergoing Implantation of Coronary Drug-Eluting Stents 3) trial is to determine the efficacy and safety of clopidogrel monotherapy compared with aspirin monotherapy beyond the standard duration of DAPT after PCI with current-generation DES in patients at high risk for recurrent ischemic events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 19 years of age
2. Patients at high risk of recurrence of ischemic events who have undergone PCI using a DES and are receiving standard DAPT (12 months* or more for myocardial infarction and 6 months* or more for non-myocardial infarction)
3. Patients at high risk for recurrent ischemic events, which were defined as one or more of the following clinical or lesion characteristics.

   A. Clinical characteristics
   1. Patients with prior myocardial infarction.
   2. Patients with diabetes mellitus who receive oral hypoglycemic agent or insulin.

   B. Complex lesion characteristics Complex lesion was defined as one or more of the following.
   1. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) and is able to assess the side branch ostium
   2. Chronic total occlusion (≥3 months) as target lesion
   3. PCI for unprotected left main disease (left main ostium, body, or distal bifurcation including non-true bifurcation lesions)
   4. Long coronary lesions (implanted stent length ≥38 mm)
   5. Multi-vessel PCI (≥ 2 vessels treated at one PCI session)
   6. Multiple stent needed (≥ 3 stents per patient)
   7. In-stent restenosis lesion as target lesion
   8. Severely calcified lesion (encircling calcium in angiography) i . Ostial lesions of left anterior descending artery, left circumflex artery, or right coronary artery
4. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.

Exclusion Criteria:

1. Known hypersensitivity or contraindications to study medications (aspirin or clopidogrel)
2. Patients who need continuous anticoagulant therapy.
3. Patients who require DAPT due to atherosclerotic disease other than coronary artery disease
4. Patients who are scheduled for revascularization treatment of coronary artery
5. A patient who are taking single antiplatelet therapy at screening
6. Pregnant or lactating women
7. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5506 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Rates of major adverse cardiac and cerebrovascular event (MACCE) | 1-year after last patient enrollment
  a composite of all-cause death, myocardial infarction, or stroke

SECONDARY OUTCOMES:
Rates of all-cause death | 1-year after last patient enrollment
  Death by any cause
Rates of cardiovascular death | 1-year after last patient enrollment
  Death by cardiovascular cause
Rates of myocardial infarction | 1-year after last patient enrollment
  Myocardial infarction
Rates of stroke | 1-year after last patient enrollment
  Stroke
Rates of stent thrombosis | 1-year after last patient enrollment
  definite or probable by Academic Research Consortium [ARC] definition
Rates of all-cause death or MI | 1-year after last patient enrollment
  A composite of all-cause death or MI
Rates of cardiovascular death or MI | 1-year after last patient enrollment
  A composite of cardiovascular death or MI
Rates of cardiovascular death, MI, or stroke | 1-year after last patient enrollment
  A composite of cardiovascular death, MI, or stroke
Rates of cardiovascular death, MI, or stent thrombosis | 1-year after last patient enrollment
  A composite of cardiovascular death, MI, or stent thrombosis
Rates of major Bleeding | 1-year after last patient enrollment
  BARC [Bleeding Academic Research Consortium] types 3 or 5
Rates of bleeding | 1-year after last patient enrollment
  BARC [Bleeding Academic Research Consortium] types 2, 3, or 5
Rates of upper gastrointestinal clinical event | 1-year after last patient enrollment
  A composite of upper gastrointestinal clinical event
Rates of gastrointestinal ulcer or bleeding | 1-year after last patient enrollment
  A composite of gastrointestinal ulcer or bleeding
New diagnosed rates of gastroesophageal reflux disease (GERD) | 1-year after last patient enrollment
  Gastroesophageal reflux disease (GERD)
Rates of NACE (Net adverse clinical events) | 1-year after last patient enrollment
  MACCE + BARC type 3 or 5 bleeding
Rates of Target-lesion revascularization (TLR) | 1-year after last patient enrollment
  Target-lesion revascularization (TLR)
Rates of Target-vessel revascularization (TVR) | 1-year after last patient enrollment
  Target-vessel revascularization (TVR)
Rates of any revascularization | 1-year after last patient enrollment
  any revascularization including TLR, TVR, and non-TVR re-percutaneous coronary intervention
Medical cost | 1-year after last patient enrollment
  Medical cost

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi KH, Park YH, Lee JY, Jeong JO, Kim CJ, Yun KH, Lee HC, Chang K, Park MW, Bae JW, Doh JH, Cho BR, Kim HY, Kim W, Kim U, Rha SW, Hong YJ, Lee HJ, Ahn SG, Kim DI, Cho JH, Her SH, Jeon DS, Han SH, Lee JB, Lee CW, Kang D, Lee JM, Park TK, Yang JH, Lee SY, Choi SH, Gwon HC, Song YB, Hahn JY; SMART-CHOICE 3 investigators. Efficacy and safety of clopidogrel versus aspirin monotherapy in patients at high risk of subsequent cardiovascular event after percutaneous coronary intervention (SMART-CHOICE 3): a randomised, open-label, multicentre trial. Lancet. 2025 Apr 12;405(10486):1252-1263. doi: 10.1016/S0140-6736(25)00449-0. Epub 2025 Mar 30. PMID 40174599